CLINICAL TRIAL: NCT03994913
Title: An Open, Multi-center Phase Ⅰ/II Clinical Study to Evaluate the Safety and Efficacy of CT032 Humanized CD19 Autologous Car T Cell Injection in Patients With Relapsed and/or Refractory Non-Hodgkin's B Cell Lymphoma
Brief Title: Clinical Trial to Evaluate CD19 CAR T (CT032) in Patients With Relapsed and/or Refractory Non-Hodgkin's B Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CARsgen Therapeutics Co., Ltd. (Industry)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT032-NHL-01
Record Dates: First submitted 2019-06-12; First posted 2019-06-21 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Refractory B-Cell Non-Hodgkin Lymphoma; Relapsed B-cell Non-Hodgkin Lymphoma
Keywords: Relapsed and/or Refractory B-cell Non-Hodgkin Lymphoma; CAR T
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-CD19-T Cells (Experimental): The subjects are enrolled into 3 dose levels cohorts in sequence.
  Interventions: Biological: CAR-CD19 T Cells

INTERVENTIONS:
Biological: CAR-CD19 T Cells — The CAR- CD19 T cells (study drug) used in this study are chimeric antigen receptor specifically expressing T cells targeting CD19.
  Fludarabine and Cyclophosphamide are used for lymphodepletion.

SUMMARY:
This is an open-label, single arm study to evaluate the safety and tolerability of treatment with CT032 CAR-CD19 T in patients with relapsed and/or refractory non-Hodgkin's B cell lymphoma (R/R B-NHL).

DETAILED DESCRIPTION:
This study is a single-arm, open label, phase I/II clinical trial to evaluate the safety, efficacy and cellular kinetics of CT032 CAR-CD19 T cells in patients with R/R B-NHL. The study is composed of two stages, Phase I stage is for dose escalation and recommendation of phase 2 dose, and Phase II stage is to verify the efficacy and safety of the dose proposed.

ELIGIBILITY:
Inclusion Criteria:

1. The subject should participate in the clinical trial voluntarily, be fully aware of and informed of this study and sign informed consent (ICF), and be willing to follow and be able to complete all trial procedures;
2. Age 18-70 years old, male or female;
3. CD 19 positive, Relapsed and/or Refractory Diffuse large B-cell lymphoma (DLBCL) and follicular lymphoma after the transformation of Relapsed and/or Refractory DLBCL subjects by histopathological and/or cytology diagnosis; At least received second-line systemic anticancer treatments containing rituximab (or other anti-CD20 drugs) and anthracene (including autologous hematopoietic stem cell transplantation) , and had progressive disease (PD) or relapse after the latest treatment.
4. The Eastern Cooperative Oncology Group (ECOG) score is 0 or 1 point;
5. The expected survival period is more than 12 weeks;
6. Having sufficient venous pathways (for leukapheresis or intravenous blood collection) and no leukapheresis contraindications;
7. At least one measurable lesion: the long axis >1.5 cm of the lymph node lesion, or the long axis >1.0 cm of the non-lymph node lesion;
8. subject has adequate organ function at screening;
9. Women of childbearing age must undergo a serum pregnancy test with negative results before screening and lymphodepletion preconditioning with fludarabine and cyclophosphamide, and are willing to use effective and reliable method of contraception for at least 1 year after T cell infusion;
10. Male subjects who have an active sex life with a woman with reproductive potential must be willing to use very effective and reliable methods of contraception for at least 1 year after T cell infusion.

Exclusion Criteria:

If the subject meets any of the following criteria, he or she cannot participate in this trial:

1. A history of severe allergies, or a history of allergies or intolerance to fludarabine, cyclophosphamide or tocilizumab, or a history of allergies or intolerance to CAR T cell cytosolic component, or a history of allergic to beta-caprolactam antibiotics;
2. Received chemotherapy, targeted therapy, radiotherapy and other anti-tumor treatment within 14 days before peripheral blood mononuclear cells (PBMCs) collection;
3. Previously received any target of CAR T treatment, or previously received CD19 targeted drug treatment;
4. Has undergone allogeneic hematopoietic stem cell transplantation; autologous stem cell transplantation was received within 12 weeks before PBMCs collection;
5. Other malignant neoplasms existed in the previous 5 years or at the same time, with the exception of breast/cervical in situ cancer, cured basal cell carcinoma and superficial bladder tumor (Ta, Tis, T1);
6. Any uncontrollable active infection, including but not limited to active TB patients
7. subjects who had received a therapeutic dose of systemic steroid drugs (prednisone >20mg/days or equivalent doses of other hormones) or other immunosuppressants within 7 days before PBMCs collection, with the exception of those who had recently or currently used inhaled steroids;
8. Known to have active autoimmune diseases, including but not limited to psoriasis, rheumatoid arthritis, etc., that need long-term immunosuppressive therapy;
9. Patients with refractory hyponatremia and/or hypokalemia;
10. Known or existing primary or metastatic central nervous system lymphoma, or any other central neurological disease or clinically significant neurological examination with abnormal results (such as seizures, cerebrovascular ischemia/hemorrhage, dementia, etc.);
11. Within 6 months prior to signing the ICF, there were any of the uncontrolled cardiovascular, cerebral vascular disease, diabetes and pulmonary embolism, or other disease at discretion of investigators that participating in this clinical trial may harm the health of the subjects;
12. Oxygen absorption before PBMCs collection to maintain blood oxygen saturation >95% (finger vein oxygen);
13. According to the investigator, any serious or uncontrollable systemic disease, systematic comorbidities, other serious concurrent diseases (such as hemophagocytic syndrome, etc.), special circumstances of the tumor may make the subjects inappropriate to enter the study or non-compliant to the protocol, or produce significant interference to correct evaluation of study drug safety, toxicity, and validity;
14. The investigators assessed that the subjects were unable or unwilling to comply with the requirements of the research protocol;
15. Major surgical operations were performed within 4 weeks of the group (the definition of major surgery is based on the 3 and 4 levels of surgery specified in the measures for the administration of clinical application of medical technology); or has not yet been fully recovered from any previous invasive operation;
16. The toxic response of previous anti-tumor therapy has not been restored to level 1 according to the Common Terminology Criteria for Adverse Events (CTCAE), except for hair loss and;
17. Having participated in any other interventional clinical trial before administration, where the last time of drug administration is within 4 weeks or less than 5 half-lives of the test drug (the longer);
18. Women who have been pregnant, prepared for pregnancy during the trial, or are breastfeeding; or women of childbearing age and fertile men who are unwilling or unable to adopt medically recognized and effective contraceptive methods throughout the study period;
19. The investigator or a relative of his staff, a subject who may have an interest in it with the investigator or his staff.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Phase Ⅰ, Safety/Tolerability: Dose-limiting toxicity (DLT) | 28 days post administration of CAR-T cells
  Dose-limiting toxicity (DLT)
Phase Ⅰ, Safety/Tolerability: Maximum tolerated dose (MTD) | 28 days post administration of CAR-T cells
  Maximum tolerated dose (MTD)
Phase Ⅰ, Safety/Tolerability: Incidence and severity of Treatment emergent adverse events (TEAE) | 28 days post administration of CAR-T cells
  Incidence and severity of Treatment emergent adverse events (TEAE)
Phase Ⅰ, Safety/Tolerability: Incidence and severity of study treatment related AE | through 2 months post administration of CAR-T cells
  Incidence and severity of AE related to study treatment
Phase Ⅰ, Safety/Tolerability: Incidence and severity of AEs of special interest (cytokine release syndrome [CRS], CART-cell-related encephalopathy syndrome [CRES]) | through 2 months post administration of CAR-T cells
  Incidence and severity of AEs of special interest (cytokine release syndrome [CRS], CART-cell-related encephalopathy syndrome [CRES])
Phase Ⅰ, Safety/Tolerability: Incidence and severity of Dose-limiting toxicity (DLT) of dose escalation experiment | 28 days after infusion
  Incidence and severity of Dose-limiting toxicity (DLT) of dose escalation experiment
Phase Ⅰ, Safety/Tolerability: Recommended Phase II Dose (RP2D) | through 2 months post administration of CAR-T cells
  Recommended Phase II Dose (RP2D)
Phase Ⅱ, Efficacy: Overall Remission Rate (ORR) | through 6 months post administration of CAR-T cells
  Overall Remission Rate (ORR) (Partial remission and complete remission rate after infusion of CT032 CAR-CD19 T cells)

SECONDARY OUTCOMES:
Phase Ⅰ, Safety/Tolerability: Incidence and severity of Treatment emergent adverse events (TEAE) | through 24 months post administration of CAR-T cells
  Incidence and severity of Treatment emergent adverse events (TEAE)
Phase Ⅰ, Safety/Tolerability: Incidence and severity of study treatment related AE | through 24 months post administration of CAR-T cells
  Incidence and severity of AE related to study treatment
Phase Ⅰ, Safety/Tolerability: Cytokine (IL-2, IL-6,IL-8,IL-10,IFN-γ,TNF-α ) concentration (pg/mL) by MSD and CBA method | through 24 months post administration of CAR-T-cells
  Cytokine (IL-2, IL-6,IL-8,IL-10,IFN-γ,TNF-α ) concentration (pg/mL) by MSD and CBA method
Phase Ⅰ: the number of copies of CAR-CD19 T cells in peripheral blood genomes by qPCR method and CAR-CD19 T cells by flow cytometry method | through 24 months post administration of CAR-T cells
  the number of copies of CAR-CD19 T cells in peripheral blood genomes by qPCR method and CAR-CD19 T cells by flow cytometry method
Phase Ⅰ, Efficacy: Overall Remission Rate (ORR) | through 24 months post administration of CAR-T cells
  Overall Remission Rate (ORR) (Partial remission and complete remission rate after infusion of CT032 CAR-CD19 T cells)
Phase Ⅱ, Efficacy: complete response (CR) rate | through 24 months post administration of CAR-T cells
  complete response (CR) rate
Phase Ⅱ, Efficacy: duration of response (DOR) | through 24 months post administration of CAR-T cells
  duration of response (DOR)
Phase Ⅱ, Efficacy: time to response (TTR) | through 24 months post administration of CAR-T cells
  time to response (TTR)
Phase Ⅱ, Efficacy: progression-free survival (PFS) | through 24 months post administration of CAR-T cells
  progression-free survival (PFS) time
Phase Ⅱ, Efficacy: overall survival (OS) | through 24 months post administration of CAR-T cells
  overall survival (OS) time
Phase Ⅱ, Safety/Tolerability: Incidence and severity of Treatment emergent adverse events (TEAE) | through 24 months post administration of CAR-T cells
  Incidence and severity of Treatment emergent adverse events (TEAE)
Incidence and severity of o study treatment related AE | through 24 months post administration of CAR-T cells
  Incidence and severity of AE related to study treatment
Phase Ⅱ, Safety/Tolerability: Incidence and severity of AEs of special interest (CRS, CRES) | through 24 months post administration of CAR-T cells
  Incidence and severity of AEs of special interest (CRS, CRES)
Phase Ⅱ, Safety/Tolerability: Cytokine (IL-2, IL-6,IL-8,IL-10,IFN-γ,TNF-α ) concentration (pg/mL) by MSD and CBA method | through 24 months post administration of CAR-T cells
  Cytokine (IL-2, IL-6,IL-8,IL-10,IFN-γ,TNF-α ) concentration (pg/mL) by MSD and CBA method
Phase Ⅱ: the number of copies of CAR-CD19 T cells in peripheral blood genomes by qPCR method and CAR-CD19 T cells by flow cytometry method | through 24 months post administration of CAR-T cells
  the number of copies of CAR-CD19 T cells in peripheral blood genomes by qPCR method and CAR-CD19 T cells by flow cytometry method

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, Dr., Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (2):
- China (2):
  - Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No